CLINICAL TRIAL: NCT07262788
Title: A Feasibility Study of Optimal Non-Pharmacological Lifestyle Modifications in People With Type 2 Diabetes (ON LiMiT)
Brief Title: A Feasibility Study of Optimal Non-Pharmacological Lifestyle Modifications in People With Type 2 Diabetes
Acronym: ON LiMiT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown); Steno Diabetes Center Odense (Other); University of Copenhagen (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jonas Salling Quist, Senior Researcher and Associate Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-77-25
Record Dates: First submitted 2025-09-11; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Obesity; Remission; Feasibility; Diet; Overweight; Lifestyle Intervention; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The feasibility study is a 52-week, 2-arm open-label randomized diet and exercise trial including 24 individuals with newly diagnosed type 2 diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CH-rich diet with exercise (Experimental): A CH-rich diet combined with an exercise programme (n=12)
  Interventions: Other: CH-rich diet with exercise
- CH-reduced diet with exercise (Experimental): A CH-redcued diet combined with an exercise programme (n=12)
  Interventions: Other: CH-reduced diet with exercise

INTERVENTIONS:
Other: CH-rich diet with exercise — After 12 weeks of following a VLCD (Phase 1), participants begin a 6-week transition (Phase 2). During this phase, they adopt a CH-rich diet, consuming 50-55% of their total energy from carbohydrates. This involves shifting gradually but structurally from formula products to regular meals. Meal boxes and formula products aligned with their assigned diet support this shift and serve as educational tools. Phase 2 also includes an exercise program consisting of two supervised 1-hour sessions and one 1-hour unsupervised high-intensity session weekly (intensity >70% peak oxygen uptake (VO2peak) and/or >7 on the Rate of Perceived Exertion scale (RPE), equivalent to 1-3 repetitions in reserve for resistance training or vigorous intensity). For the next 34 weeks (Phase 3), participants receive ongoing diet and exercise support while purchasing and preparing their own meals according to their assigned diet. They continue with two supervised and one unsupervised group session per week.
  Arms: CH-rich diet with exercise
Other: CH-reduced diet with exercise — After 12 weeks of following a VLCD (Phase1), participants begin a six-week transition (Phase 2 ). During this phase, they adopt a CH-reduced diet, consuming 25-30% of their total energy from carbohydrates. This involves shifting gradually but structurally from formula products to regular meals. Meal boxes and formula products aligned with their assigned diet support this shift and serve as educational tools. Phase 2 also includes an exercise program consisting of two supervised 1-hour sessions and one 1-hour unsupervised high-intensity session weekly (intensity >70% peak oxygen uptake (VO2peak) and/or >7 on the RPE scale, equivalent to 1-3 repetitions in reserve for resistance training or vigorous intensity). For the next 34 weeks (Phase 3), participants receive ongoing diet and exercise support while purchasing and preparing their own meals according to their assigned diet. They continue with two supervised and one unsupervised group session peer week.
  Arms: CH-reduced diet with exercise

SUMMARY:
The overall aim of this study is to examine the feasibility of a 12-month, two-arm lifestyle intervention to induce and maintain remission of type 2 diabetes (T2D). The findings from the feasibility study will inform the recruitment, design and delivery of the interventions in a 5-arm, 24-month randomised controlled trial.

DETAILED DESCRIPTION:
Studies on T2D remission have reported varying rates of remission, often around 50% in intervention groups. These studies typically involve individuals with a recent T2D diagnosis, usually within six to ten years of diagnosis, with intervention periods most commonly lasting between twelve and twenty-four months, though durations have ranged from six to sixty months. Lifestyle interventions combining dietary changes and increased physical activity generally yield modest remission rates, but maintaining adherence over time remains challenging. Trials that include an initial phase of a very low-calorie diet, followed by ongoing structured support, tend to report higher remission rates. This emphasizes the critical role of significant and sustained weight loss. However, the most effective combination of dietary, exercise, and behavioral support strategies remains to be determined.

In addition to calorie restriction, changes in dietary composition may influence the underlying mechanisms of T2D. For instance, reducing carbohydrate intake can promote ketone production, affecting liver glucose production and improving glycemic control. Higher protein intake has been linked to an improved insulin response. Replacing saturated fats with polyunsaturated fats and increasing dietary fiber may also support glucose metabolism. However, it remains unclear whether carbohydrate-reduced or carbohydrate-rich diets are more effective in supporting long-term remission following initial weight loss.

Physical activity, particularly high-intensity exercise, plays a key role in reducing the risk of T2D, supporting weight management, and improving remission rates when combined with dietary interventions. Significant improvements in blood glucose control are usually seen with regular moderate-to-high-intensity exercise.

Moreover, there is considerable variation-or sometimes an absence-in the inclusion of key lifestyle intervention components, such as specific dietary and exercise protocols, as well as levels of supportive activities. This inconsistency complicates effective care provision for healthcare professionals and makes it difficult for individuals with T2D to adhere to non-pharmacological management recommendations.

Despite the known benefits of lifestyle modifications, initiating and maintaining these changes is challenging due to barriers such as a lack of support, motivation, and knowledge about nutrition and portion sizes. Involving individuals with T2D in designing and evaluating interventions may improve adherence, reduce participant burden, and increase the feasibility and scalability of lifestyle programs for wider implementation.

The overall aim of this study is to examine the feasibility of a 12-month, two-arm intervention designed to induce and maintain remission of T2D. After baseline measurements, participants will be randomized to one of two groups: Group A: Very-low-calorie-diet (VLCD)/weight loss followed by a carbohydrate-reduced (CH-reduced) diet combined with high-intensity exercise. Group B: VLCD/weight loss followed by a carbohydrate-rich (CH-rich) diet combined with high-intensity exercise. Participants will be blinded to the intervention arm during the VLCD phase. To determine the optimal macronutrient composition of the Mixed Meal Tolerance Test (MMTT) for subsequent testing, participants will attend three MMTTs in random order at baseline. The MMTTs consists of three different macronutrient compositions (X energy percentage (E%)carbohydrate, XE% protein, XE% fat; XE% carbohydrate, XE% protein, XE%fat; E% carbohydrate, XE% protein, XE% fat)

Feasibility will be evaluated based on the recruitment process, intervention acceptability, and participant adherence. This includes assessing whether the intervention components and outcome measurements are delivered and conducted as intended. Additionally, the study will examine how these elements perform in a real-life setting among individuals with T2D. Findings from this feasibility study will inform recruitment strategies, study design, and implementation of a subsequent five-arm, 24-month randomized controlled trial.

Specific aims:

1. To study the recruitment process (including recruitment of general practitioners and participants) and identify related barriers and facilitators.
2. To investigate retention, adherence, and acceptability of the interventions (carbohydrate-reduced or carbohydrate-rich diet combined with high-intensity exercise), including participant experiences with the intervention components and data collection procedures.
3. To assess whether the intervention is delivered as intended, covering supervised/unsupervised sessions, study visits, online support, and group education.
4. To evaluate the effectiveness of safety procedures in responding to changes in participants' glycemic control, blood pressure, physical injuries, and related risk markers.
5. To determine the optimal macronutrient composition and sampling schedule for the Mixed Meal Tolerance Test (MMTT).
6. To explore the potential impact of the two interventions on T2D remission rates and related metabolic outcomes such as body weight, body composition, blood pressure, vascular function, glycemic control, lipid profile, beta-cell function, and inflammation.

ELIGIBILITY:
Building on previous findings from T2D remission studies involving VLCD interventions, the study include individuals with recently diagnosed T2D who are overweight or obese and not receiving insulin therapy. This subgroup has demonstrated the greatest benefit from significant weight loss. Participants using GLP-1 receptor agonists (GLP-1 RAs) are eligible, provided their weight has been stable for at least three months prior to inclusion. Individuals on insulin therapy will be excluded. Allowing GLP-1 RA use enhances the study's generalizability, as approximately 29% of people with T2D in Denmark are currently treated with these medications.

Inclusion Criteria:

* Diagnosis of T2D and treatment with lifestyle and/or oral anti-diabetic medication and/or glucagon-like peptide-1 receptor agonists (GLP-1RAs)
* HbA1c between 36-86 mmol/mol
* T2D duration of ≤6 years
* BMI ≥27 kg/m2
* Body weight changes over 3 months ≤3 kg

Exclusion Criteria:

* Insulin treatment within 6 months prior to screening (any type)
* Heart failure (ejection fraction<40%) and treated with SGLT-2i (current or planned)
* Kidney disease (eGFR<60 ml/min) and treated with SGLT-2i (current or planned)
* Physical comorbidity, which precludes the physical activity during intervention
* Dietary restrictions or allergies making the participant unable adhere to the dietary interventions
* Unable to comply with trial procedures and/or interventions
* Alcohol/drug abuse
* Planned or present pregnancy
* Unstable psychiatric disease
* Diagnosed with binge eating disorder
* Participation (present or planned) in other clinical trials including lifestyle or pharmacy trials for any condition
* If HbA1c ≥60 mmol/mol and the participant is on 2 or more anti-diabetic drugs a positive GAD65 and/or stimulated C-peptide <800 pM excludes the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility testing of diet adherence | Baseline, week 18, 24, 36 and 52.
  Derived from myfood24 dietary recalls collected over three consecutive days at pre-specified time points. A recall day is adherent if E% carbohydrate is within the arm-specific target ±10 E%. Participant-level percent compliance at each time point is calculated as (adherent recall days / valid recall days) × 100.
Feasibility testing of exercise adherence | 3 sessions pr. week, from week 13 to 52.
  Adherence is assessed based on self-report and measured (wearable heart rate monitor) using study-app and calculated as number of completed sessions / total prescribed sessions.
Feasibility testing of GP recruitment & safety procedures - quantitative assessment | Through study completion, an average of 52 weeks.
  The recruitment of GPs will be assessed based on the number who express interest, attend instruction and sign collaboration agreements. The reasons for GP non-participation or withdrawal will be documented and, if possible, the GPs will be interviewed. Contacts with GPs that are safety-related, and their responses, including the outcomes of medication changes, will be recorded.
Feasibility testing of GP experiences and study procedures - qualitative assessment | Through study completion, an average of 52 weeks.
  Interviews with with one GP or staff member from each participating clinic will explore experiences with study procedures, including barriers and opportunities related to recruitment and medication discontinuation, as well as any unintended consequences.
Feasibility testing of participant recruitment & retention | Through study completion, an average of 52 weeks.
  Registered numbers of: individuals expressing interest in the project, participants completing pre-screening (telephone interview) and in-person screening, participants included in the study, drop-outs and completers. Reasons for exclusion or withdrawal will be documented.
Feasibility testing of intervention participation - quantitative assessment | Through study completion, an average of 52 weeks.
  The degree of implementation of intervention activities and the extent of participant engagement will be measured by tracking attendance and completion of planned intervention components, including intervention visits, supervised and unsupervised exercise sessions, phone calls, at-home measurements, group-based education sessions, and peer support activities. Data will be collected via REDCap (8.10.18, Vanderbilt University, TN, USA) and study logs to quantify the proportion of completed versus scheduled ac-tivities for each participant.
Feasibility testing of intervention participation - qualitative assessment | Through study completion, an average of 52 weeks.
  Group-based diet and exercise sessions will be observed to assess how the intervention is delivered in practice and how participants engage with the activities. Field notes will document group dynamics, adherence to session protocols, and contextual factors. Field notes will also inform interview guides and supplement interview data.
Feasibility testing of protocol adherence - number of days with deviations | Through study completion, an average of 52 weeks.
  Total number of days during which participants did not adhere to the planned intervention protocol or experienced protocol devia-tions during the three intervention phases.
Feasibility testing of acceptability and experiences | Through study completion, an average of 52 weeks plus a 3-month follow-up interview with participants.
  Interviews with participants, dieticians and exercise instructors.

SECONDARY OUTCOMES:
Evaluation of dietary screener to assess adherence | Every 2 weeks from week 15 to week 52.
  A dietary screener will be used to generate a binary off-track flag to enable timely dietitian outreach when participants may need support to improve adherence during the study period. As part of the dietary screener, participants will complete an overall self-assessment of adherence to their allocated diet during the past 7 days. Participant ratings will be compared with the dietitian's adherence rating following flagged checks, and interrater agreement (participant vs. dietitian) and agreement with MyFood24-derived adherence will be explored.
Dietary intake | Measured at baseline, week 18, 24, 36 and 52.
  Dietary intake, including energy intake (kcal/day) and macronutrient intake (total in grams and E% per day) and micronutrient intake (units/day) intake based on 3-days' dietary recalls based on MyFood24.
Diabetes remission | Measured at week 12, 18 and 52.
  Number of participants with HbA1c < 48 mmol/mol without diabetes medication.
Body weight (kg) | Changes from baseline to the end of the intervention measured at four time points (baseline, week 12, 18 and 52).
  Measured to nearest 0.1 kg using a digital scale. Fasted state.
Achieved clinically relevant weight loss (≥10%) | Measured at baseline, week 12, 18 and 52.
  Number of participants who achieved a weight loss of at least 10% of their baseline body weight. Measured to nearest 0.1 kg using a digital scale. Fasted state.
HbA1c (mmol/mol and %) | Measured at screening, baseline, week 12, 18, 30, 42 and 52.
  Assessed from blood samples collected in non-fasting state.
GAD65 Antibodies (U/mL) | Measured at screening.
  Assessed from blood samples collected in non-fasting state.
Proinsulin (pmol/L) | Measured at screening.
  Assessed from blood samples collected in non-fasting state.
Blood lipids (mmol/L) | Measured at baseline, week 12, 18 and 52.
  Fasting concentrations of: Total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides.
Marker of kidney function - eGFR (mL/min) | Measured at baseline, week 12, 18 and 52.
  Estimated glomerular filtration rate (eGFR).
Marker of kidney function - Creatinine (μmol/L) | Measured at baseline, week 12, 18 and 52.
  Concentration of creatinine, assessed from blood sample in fasting state.
Marker of kidney function - Potassium (mmol/L) | Measured at baseline, week 12, 18 and 52.
  Concentration of potassium, assessed from blood sample in fasting state.
Marker of kidney function - Sodium (mmol/L) | Measured at baseline, week 12, 18 and 52.
  Concentration of sodium, assessed from blood sample in fasting state.
Plasma Albumin (g/L) | Measured at baseline, week 12, 18 and 52.
  Fasting concentration of plasma albumin.
Plasma Hemoglobin (g/L) | Measured at baseline, week 12, 18 and 52.
  Fasting concentration of plasma hemoglobin.
White Blood Cells (10⁹/L) | Measured at baseline, week 12, 18 and 52.
  Fasting concentration of white blood cells.
Height (m) | Measured at baseline.
  Measured using a using an ultrasonic device to nearest 0.1 cm in order to calculate BMI.
Body weight (kg) | Measured at week 11, 12, 16, 18, 51 and 52.
  Measured to nearest 0.1 kg, in the morning, after urinating, before ad libitum diet acc to ad libitum intake of allocated intervention diet, using wireless scales at participants' home.
Body mass index (kg/m^2) | Measured at baseline, week 12, 18 and 52.
  Calculated from body weight (kg) and height (m). Fasted state.
Gut Microbiome Composition | Collected at baseline, week 12, 18 and 52.
  Fecal samples will be analyzed for microbiome composition and diversity using 16S rRNA gene sequencing and shotgun metagenomic sequencing.
Urine spot samples for dietary biomarkers (home collection) | Collected at week 18 and 52.
  Participants will collect three consecutive morning midstream urine samples and four additional spot urine samples at home. Urine samples will be analyzed by metabolomic profiling to quantify urinary concentrations of at least 10 dietary biomarkers, including Sulforaphane-N-acetylcysteine (broccoli), Proline betaine (citrus fruits), Carnosine (meat), and 3,5-dihydroxybenzoic acid glucuronides (whole grains).
Urine Albumin-to-Creatinine Ratio (at site) | Measured at baseline, week 12, 18 and 52.
  Urine spot samples will be collected to assess renal function and diabetes-related kidney involvement.
Saliva microbiome composition | Collected at baseline, week 12, 18 and 52.
  Saliva samples, analyzed for microbial composition changes via 16S rRNA and metagenomic.
Metabolites - MMTT | Measured at baseline, week 12, 18 and 52.
  Concentrations of metabolites, including but not limited to: glucose, triglycerides, free fatty acids (FFA), glycerol, fasting lipoproteins, intact and split proinsulin, C-peptide and alanine, measured in response to high-carbohydrate versus high-protein isocaloric liquid meals. Blood samples will be collected at 8 time points: fasting (-10 and 0 minutes) and postprandially at 30, 60, 90, 120, 180, and 240 minutes during the MMTT.
Hormones and other blood analyses during MMTT | Measured at baseline, week 12, 18 and 52.
  Concentrations of hormones involved in glucose and lipid metabolism and appetite regulation, may include but not limited to: insulin, glucagon, C-peptide, GLP-1, GIP, ghrelin, PYY, CCK, FGF21, GDF15, LEAP2. Blood samples will be taken at 8 measurements points: at fasting (-10 and 0 minutes) and postprandially at 30, 60, 90, 120, 180, and 240 minutes during the MMTT.
Subjective appetite sensations | Measured at baseline, week 12, 18 and 52.
  Rated using visual analogue scales (VAS) and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, or sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before". VAS are collected at multiple timepoints during MMTT: at -25 to -10 minutes (pre-meal baseline), and at 70-85, 160-175, and 220-235 minutes post-meal.
Physical activity | Measured at baseline, week 12, 18 and 52.
  Physical activity (PA) including but limited to: PA (time spent at different intensities (sedentary activity, low light activity, high light activity, moderate to vigorous activity, vigorous activity), PA (total counts, counts/min), PA energy expenditure (kcal/day), PA (MET hours) and timing of PA (hh:mm) will be objectively assessed using a thigh-mounted accelerometer (SENS Motion). Participants will wear the device 24 hours/day for 10 consecutive days prior to visits. Data will provide time-stamped estimates of sedentary time, time spent standing, walking, bicycling, and intensity of movement.
Waist circumference (cm) | Measured at baseline, week 12, 18 and 52.
  Measured using tape measure to the nearest 0.5 cm. Fasted state.
Hip circumference (cm) | Measured at baseline, week 12, 18 and 52.
  Measured using tape measure. Fasted state.
Waist/hip ratio | Measured at baseline, week 12, 18 and 52.
  The ratio of the circumference of the waist to that of the hips.
Fat mass (kg) | Measured at baseline, week 12, 18 and 52.
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Fat free mass (kg) | Measured at baseline, week 12, 18 and 52.
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Fat percentage (%) | Measured at baseline, week 12, 18 and 52.
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Bone mass (kg) | Measured at baseline, week 12, 18 and 52.
  Measured by Dual-energy X-ray Absorptiometry in a fasted state.
Marker of liver function - Degree of liver fibrosis (kPa) | Measured at baseline, week 12, 18 and 52.
  Measured by FibroScan in a fasted state.
Marker of liver function - Degree of liver steatosis (dB/m) | Measured at baseline, week 12, 18 and 52.
  Measured by FibroScan in a fasted state.
Marker of liver function - FIB-4 Index | Measured at baseline, week 12, 18 and 52.
  Will be calculated from participants' age and fasting concentration of aspartate-aminotransferase (U/L), alanine-aminotransferase (U/L) and thrombocytes (x10^9/L).
Cognition | Measured at baseline, week 12 and 52.
  Cognitive functions will be assessed by Screen for Cognitive Impairment in Psychiatry Danish Version (SCIP-D) together with the Trail Making Test-Part B (psychomotor speed and executive function).
Food choice - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT). Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Food attention - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Measured using eye tracking in response to looking at food pictures during Steno Biometric Food Preference Task (SBFPT). Includes the following parameters: Gaze: Time spent (ms and %) and visits (n); and fixations: Time to first fixation (ms), time spent (ms and %), fixation count (n), first fixation duration (ms), average fixation duration (ms). Distance to screen (mm), and gaze direction bias (ratio) which is calculated as the number of trials in which the first fixation was directed to a food image as a proportion to all trials. A bias score #0.5 indicates attention towards one food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates attention towards the other food images.
Food reaction time (ms) - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Reaction time during forced food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fatsavoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT).
Explicit liking - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savouryand low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT). Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this foodright now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Implicit wanting - Food preferences and food reward | Measured at baseline and test visits at week 12, 18 and 52 (T=-60 min and T=120 min).
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT). Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time (a frequency-weighted algorithm). In this frequency-weighted algorithm a positive score indicates a morerapid preference for a food type over another food type and a negative score indicates the opposite. A score of zero indicates that food types are equally preferred. The frequency weighted algorithm isused so the implicit wanting score is influenced by both selection (positively contributing to the score) and non-selection (negatively contributing to the score) of food type. Scores for implicit wanting typically range from -100-100 (due to reaction time there is no fixedmin-max value).
Explicit wanting - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT). Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Unspecified exploratory outcome - Food preferences and food reward | Measured at baseline, week 12, 18 and 52.
  Unspecified exploratory outcomes related to the 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the Steno Biometric Food Preference Task (SBFPT).
Systolic blood pressure (mmHg) | Measured at baseline, week 12, 18 and 52.
  Measured under resting and fasting conditions.
Diastolic blood pressure (mmHg) | Measured at baseline, week 12, 18 and 52.
  Measured under resting and fasting conditions.
Resting heart rate (bpm) | Measured at baseline, week 12, 18 and 52.
  Measured in a fasted and rest state.
Cardiac rhythm (ECG) | Measured at baseline.
  A standard 12-lead resting ECG will be performed to assess cardiac rhythm and detect potential contraindications for maximal exercise testing. This screening is conducted to ensure participant safety prior to performing the VO₂peak test.
Peak oxygen uptake (ml O2/min) | Measured at baseline, week 12, 18 and 52.
  Peak oxygen consumption (VO2peak) as a measure of cardiorespiratory fitness will be measured by an incremental bicycle ergometer test.
Cardiorespiratory fitness (ml O2/min/kg) | Measured at baseline, week 12, 18 and 52.
  Peak oxygen consumption (VO2peak) per kg body weight as a measure of cardiorespiratory fitness. Measured by an incremental bicycle ergometer test.
Time-in-range (% 3.9-10.0 mmol/L) | Measured at baseline, week -1 and 51.
  Measured using a blinded continuous glucose monitoring device (CGM). The sensor will be placed subcutaneously on the upper arm or abdomen, and worn for 10-14 days prior to visits.
Time-below-range (% <3.9 mmol/L) | Measured at baseline, week -1 and 51.
  Measured using a blinded continuous glucose monitoring device (CGM). The sensor will be placed subcutaneously on the upper arm or abdomen, and worn for 10-14 days prior to visits.
Time-above-range (% >10.0 mmol/L) | Measured at baseline, week -1 and 51.
  Measured using a blinded continuous glucose monitoring device (CGM). The sensor will be placed subcutaneously on the upper arm or abdomen, and worn for 10-14 days prior to visits.
Coefficient of variation (CV) of glucose concentrations | Measured at baseline, week -1 and 51.
  Measured using a blinded continuous glucose monitoring device (CGM). The sensor will be placed subcutaneously on the upper arm or abdomen, and worn for 10-14 days prior to visits.
Heart rate (bmp) | Measured from weeks 16 to 51 during exercise sessions.
  Assessed from GPS-based smart watch.
Self-reported quality of life | Measured at baseline, week 12 and 52.
  Assessed using the Quality of Life (12-Item Short Form Survey, SF-12), which measures health-related quality of life across physical and mental health domains. The questionnaire includes 12 items and yields two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Scores range from 0 to 100, with higher scores indicating better health status. A PCS score of 50 or below may indicate physical health impairment, while an MCS score of 42 or below may suggest clinical depression.
Self-reported health-related quality of life | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire European Quality of Life - 5 Dimensions (EQ-5D). EQ-5D comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on 3 or 5 levels of severity. A health utility index score is derived, ranging from values below 0 (where 0 represents death and negative values represent states worse than death) to 1 (full health). Higher scores indicate better health-related quality of life.
Changes in sum score The 25-item Bodily Distress Syndromes (BDS) checklist | Measured at baseline, week 12 and 52.
  Measure of severity of symptom burden. The number of non-missing (answered) items in the 25-item Bodily Distress Syndromes (BDS) checklist (from bds1 to bds25) is counted for each individual to determine if enough data is available to compute a score. Then, if at least 13 items are answered, the average of the available responses is calculated, scaled to a 0-100 range, rounded to the nearest whole number, and saved as the BDS sum score. Lower value is better.
Changes in symptom cases | Measured at baseline, week 12 and 52.
  For each of the following domains: cardiopulmonary symptoms (b1-b6), gastrointestinal symptoms (b7-b13), musculoskeletal symptoms (b14-b20) and general symptoms (b21-b25).Bimodal variable for cases - Number of symptoms scored above 1 (including Somewhat, Quite a bit & A lot). Participants reporting ≥4 such symptoms and with fewer than 3 missing responses will be classified as a case being at least four symptoms within each domain (binary variable: 1 = case, 0 = non-case).
Self-reported diabetes distress | Measured at baseline, week 12 and 52.
  Assessed from the Problem Areas in Diabetes Scale (PAID-5 scale) comprising five of the emotional-distress questions of the full PAID items. Each item can be rated from 0 to 4. A total score of ≥ 8 indicates possible diabetes related emotional distress.
Self-reported loneliness | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire The Three Item Loneliness Scale (TILS). TILS consists of 3 items assessing subjective feelings of loneliness and social isolation. Scores range from 3 to 9, with higher scores indicating greater loneliness. A score of 6 or above has been used as a cut-off to indicate elevated loneliness in population-based studies.
Self-reported sleep quality | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire Pittsburgh Sleep Quality Index. The questionnaire consists of 19 items. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Self-reported self-efficacy for nutrition change | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire Self-efficacy for nutrition change (SEFNC). SEFNC assesses individuals' confidence in their ability to maintain healthy eating habits in challenging situations over the next six months. The scale includes 9 items addressing common barriers such as emotional distress, lack of support, time pressure, and disrupted routines. Each item is rated on a percentage scale from 0% ("Not at all confident") to 100% ("Completely confident"), in 10% increments. A higher mean score indicates greater self-efficacy for sustaining nutrition-related behavior change.
Self-reported social support for eating habits | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire Social Support for Eating Habits Questionnaire. The questionnaire includes 10 items rated separately for family and friends, assessing both supportive and unsupportive behaviors related to dietary change. Items are rated on a scale from 1 (Not at all) to 5 (Very often), with 8 indicating "Not applicable." Higher scores on supportive items reflect greater perceived support; higher scores on unsupportive items reflect greater social barriers.
Self-reported food addiction | Measured at baseline, week 12 and 52.
  Assessed from the questionnaire Yale food addiction scale (YFAS). It consists of 25 items evaluating symptoms such as loss of control over eating, continued use despite negative consequences, and withdrawal. The scale provides both a symptom count score (ranging from 0 to 11) and a diagnostic threshold indicating the presence of food addiction. Higher scores indicate more severe food addiction symptomatology. A diagnosis is assigned if a certain number of symptoms are endorsed along with clinically significant impairment or distress
Adverse event | Through study completion, an average of 52 weeks.
  Number and description of adverse events and serious adverse events reported during the intervention period.
Exercise intensity (%VO2peak) | Measured at baseline, week 12, 18 and 52.
  Heart rate assessed from GPS-based smart watch and corresponding %VO2peak (measured at test visits).
Exercise intensity (Rate of Perceived Exertion Scale) | 3 sessions pr. week, from week 13 to week 52.
  Rate of perceived Exertion on a 0 to 10 scale (0 being no exertion at all and 10 being a maximum effort).
Cardiac index - MMTT | Measured at baseline, week 12, 18 and 52.
  Cardiac Index (L/min/m²) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Cardiac output - MMTT | Measured at baseline, week 12, 18 and 52.
  Cardiac output (L/min) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Systemic vascular resistance - MMTT | Measured at baseline, week 12, 18 and 52.
  Systemic vascular resistance (dyn*s/cm5) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Stroke volume index - MMTT | Measured at baseline, week 12, 18 and 52.
  Stroke volume index ( mL/m2) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Heart rate variability - MMTT | Measured at baseline, week 12, 18 and 52.
  Heart rate variability (ms) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Heart rate - MMTT | Measured at baseline, week 12, 18 and 52.
  Heart rate (bmp) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Blood pressure - MMTT | Measured at baseline, week 12, 18 and 52.
  Blood pressure (mmHg) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Blood pressure variability - MMTT | Measured at baseline, week 12, 18 and 52.
  Blood pressure variability (mmHg) will be measured using the non-invasive Finapres Nova device at -40 min for 12 min (pre-meal baseline), and at 10, 30, 60, 90, 120, 180, 240 for 8 min during the MMTT.
Timing - sleep pattern | Measured from week 16 - 51 (GSP-based smart watch) and at baseline, week 12, 18 and 52 (SENS Motion).
  Sleep timing (hh:mm) will be measured with a GPS-based smartwatch and a thigh-mounted accelerometer (SENS Motion).
Duration - sleep pattern | Measured from week 16 - 51 (GSP-based smart watch) and at baseline, week 12, 18 and 52 (SENS Motion).
  Sleep duration (minutes) will be measured with a GPS-based smartwatch and a thigh-mounted accelerometer (SENS Motion).
Variability - sleep pattern | Measured from week 16 - 51 (GSP-based smart watch) and at baseline, week 12, 18 and 52 (SENS Motion).
  Sleep variability (minutes) will be measured with a GPS-based smartwatch and a thigh-mounted accelerometer (SENS Motion).
Efficiency - sleep pattern | Measured from week 16 - 51 (GSP-based smart watch) and at baseline, week 12, 18 and 52 (SENS Motion).
  Sleep efficiency (%) will be measured with a GPS-based smartwatch and a thigh-mounted accelerometer (SENS Motion).
Wakefulness - sleep pattern | Measured from week 16 - 51 (GSP-based smart watch) and at baseline, week 12, 18 and 52 (SENS Motion).
  Sleep wakefulness (%) will be measured with a GPS-based smartwatch and a thigh-mounted accelerometer (SENS Motion).

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Salling Quist Senior Researcher and Associate Professor, PhD, Principal Investigator — Steno Diabetes Center Copenhagen, University of Copenhagen - Department of Biomedical Sciences
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No